CLINICAL TRIAL: NCT05121454
Title: Validation of an Automatic Continuous Urine Output (CUO) and Intra-Abdominal Pressure (IAP) Measuring Device
Brief Title: Validation of Serenno CUO and IAP Measuring Device
Status: Completed | Type: Observational
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Principal Investigator, Barak Cohen, MD, Vice Chair Division of Anesthesiology, Intensive Care Medicine and Pain management, Tel-Aviv Medical Center, Sackler faculty of medicine, Tel-Aviv University, Israel, Tel-Aviv Sourasky Medical Center
Other Study IDs: 0406-21-TLV
Record Dates: First submitted 2021-10-31; First posted 2021-11-16 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Urinary Catheter; Laparoscopic Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Serenno Sentinel, model Alpha 2.0, software version: 8.0 — intra-abdominal pressure measurements compared to a Foley Manometer at different insufflation pressures between 5 and 25 cmH20 at 30seconds intervals.

SUMMARY:
Serenno Medical Automatic Urine Output measuring device is intended to measure volumetric flow rate (total volume and rate) of urine produced per minute over long periods by a patient with a urinary catheter as well as high resolution IAP via bladder pressure (IBP). The device comprises a control unit located near the bed, and a disposable unit connected between the catheter and the urine collection tube/bag. The disposable unit is connected to the control unit with a tube.

Frequent and accurate Intra-Abdominal Pressure measurements facilitate management of critical care patients, yet this parameter is normally measured manually, intermittently, and inaccurately. Automating IAP measurement will increase responsiveness, reduce workload, and potentially improve outcomes. The investigators goal is to validate the accuracy urinary catheter estimates of IAP compared to the gold standard during the application of a wide range of pressures controlled by a validated closed-loop insufflation reference.

Primary Objective:

The study objective is to evaluate the accuracy of the Serenno Medical IAP measurements in patients with indwelling urinary catheters vs. the gold standard - the Foley Manometer

DETAILED DESCRIPTION:
The system which is the subject of the current study comprises two connected parts, the controller and the disposable.The disposable is a special pressure sensing fluid pump connected serially between the catheter and urine bag. The pump is operated by controlled air pressures sent via three tubes from the controller. The pump operates in strokes, with each stroke passing exactly 1ml of fluid from the input port which is connected to the catheter in the patients' bladder, to the output port, which is connected via a long tube to the urine collection container (bag or other). Since each stroke of the pump is known and constant, and the monitor is counting and timing the strokes both current urine production rate, flow rate and cumulative urine volume over any period can be measured. The pump is also unique in that its design allows the controller to measure the fluid pressure at both the input port, as well as in the output port allowing automatic high resolution Intra-Abdominal pressure monitoring in parallel and without interrupting the Urine Output monitoring.

Ongoing pressure monitoring and supporting algorithm remove the need to manually fill and empty the bladder and avoid interrupting urine output monitoring. The method also delivers multiple per-hour IAP measurements and is able to show trends to correlate to patient angle and condition.

Urine pumping eliminates all problems associated with existing systems and methods for measuring urine output. The volume measurement is accurate since it is measured in a "digital" format, by calculating of number of fixed bolus units transferred. Dependent loop and tube related accumulation are avoided since the pump passes a fixed volume of urine, no matter how it is distributed in the drain tube. Similarly, urine composition, temperature, production rate, specific weight are irrelevant to the pumping accuracy, as well as patient/bed motions and vibrations.

The controller operates the pump in a cyclic fashion. First, it measures the urine pressure inside the patients' bladder, as it is expressed as the pressure in the pump input port. A positive pressure of a few mmHg indicates that there is a minimal volume of urine in the bladder (and also indicate IAP). The controller then runs the pump for a single cycle, removing 1cc of urine from the bladder and repeating the pressure measurement and pump operation until the pressure at the input port drops back to zero - indicating an empty bladder, then stops. This process repeats for the duration of use. UO is calculated by the number of cycles and time of each divided by the relevant timeframe, normally cc/h.Providing a continuous fully automated and accurate method to measure IAP could be important in several clinical setups. Current reference methods for IAP measurement are intermittent and cumbersome. They are affected by body position, zero reference, and highly user dependent.

Study design allows a large range of pressure levels assessed simultaneously between the study device and the gold standard.

The study population is a good representation of the target population, being sedated in the supine position.

Subjects will be recruited in the pre-operative period by the study staff. b. Study Duration (per subject and total):

33 patients (3 pilot patients) Durations from study device connection to removal during the OR procedure. Estimated 15 minutes.

Total study duration is estimated as 12 months from its initiation. c. Study procedure: Screening Subjects will be screened according to eligibility criteria. The investigator will explain to the patient the nature of the study, its purpose, the procedures involved, the expected duration, the potential risks and benefits involved and any discomfort it may entail. The patients will be informed that participation in the study is voluntary, that the participants may withdraw from the study at any time and that withdrawal of consent will not affect his/her subsequent medical treatment (if any) or relationship with the treating physician.

System set up, initiate data collection and follow up.

A sealed envelope containing a set of 5 computer-generated random pressure insufflation targets will be opened. This will be used for stage 9.

A new and sterile study device disposable pump will be used for each patient (study device).

A new and sterile IAP Foley Manometer will be used for each patient. The Foley Manometer will be positioned so it is visible, stationary and it's zero point is at the same level as required in the device installation requirements at the level of the bladder.

The study device Controller unit will be cleaned per OR procedures between uses (study device).

If catheter is installed in the OR (as part of the OR requirements) it should not be drained to a bag and immediately connected to the Foley Manometer The investigator or study staff in the OR will connect the study device and IAP Foley Manometer to the patient urine line, noting the date and time.

If needed for the IAP Foley Manometer reading and/or study device a fluid bolus of 25cc will be introduced and recorded.

If needed, the battery of the device will be replaced as needed. Data storage card from the device will be backed up between uses.

An investigator or study staff will perform a series of intermittent measurements using the Foley Manometer (manual IAP measurement) while the surgeon is changing the insufflation pressures to the preselected random targets, all between 8-25 mmHg. Each level will be maintained for a duration of 30 seconds.

The study device will measure and save ongoing IAP during the process, measurements gathered by the study device will not be visible once measurements have started and can only be retrieved from the device memory during analysis. Urine Output functions will be turned off.

After the set of measurements, the study device disposable unit and the manometer unit will be disconnectedNote: Disconnection of the patient from the study device control unit is considered as study termination.

The surgical procedure will resume as normal.

Study termination: system removal and documentation

1. The investigator in the OR will disconnect the study device and IAP Foley Manometer from the patient urine line.
2. The disconnected equipment will be sealed in a bio-hazard bag marked with the subject study number and returned to Serenno as soon as possible. After inspection it will be destroyed at the responsibility of Serenno.
3. The SD card carrying the patients' data will be removed from the controller, marked with the subject study number,. A new, blank SD card will be inserted in the controller in preparation for the next patient.
4. The controller can be used with the next patient after cleaning and disinfection per the OR normal operating procedures and IFU (instruction for use).
5. Patients' CRF will include information covering the study period will be extracted from the patient's medical files. The data included in the CRF shall include, at a minimum: i. Hospital records,, weight, BMI, ASA score or equivalent at admission. ii. The set of Foley Manometer IAP measurements and the set of insufflation levels and their timing preformed during the procedure (corresponding to the random values from the envelope).

iii. Record of any unusual events during the study period, made by the OR staff iv. Record of any unusual events during the study period, made by a technical representative.

v. Control unit and disposable units serial numbers used per session

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients aged 18 years or more.
2. Patients scheduled for laparoscopic surgical procedure requiring an indwelling urinary catheter.
3. Providing informed consent.

Exclusion Criteria:

1. Known urological pathology
2. Known pregnancy
3. Cognitive and/or psychiatric impairment precluding informed consent.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients undergoing laparoscopic surgical procedure requiring an indwelling urinary catheter.
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2021-11-15 (Actual); Primary Completion 2022-03-07 (Actual); Study Completion 2022-03-07 (Actual)

PRIMARY OUTCOMES:
Accuracy of intra-abdominal pressure measurements according to the study device | 10 minutes prior to surgery
  Intra-abdominal pressure in mmHg compared to measurements from a Foley Manometer at different insufflation pressures between 8 and 25 cmH20 at 30-seconds intervals.

CONTACTS AND LOCATIONS:
Overall Officials: Barak Cohen, MD, Principal Investigator — Vice Chair Division of Anesthesiology, Intensive Care Medicine and Pain management
Locations (1):
- Division of Anaesthesia, Intensive Care, and Pain Management, Tel-Aviv Medical Center, Tel Aviv, Israel